CLINICAL TRIAL: NCT05431855
Title: Self-management of HIV and Alcohol Reaching Emerging Adults: Project Engage
Brief Title: Project Engage: A Wrist Biosensor-based mHealth Suite to Support Alcohol Intervention in Young People Living With HIV
Acronym: SHARE Engage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: University of Florida (Other); University of Michigan (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Sylvie Naar, Distinguished Endowed Professor, Florida State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00002534; 1P01AA029547-01 (NIH)
Record Dates: First submitted 2022-06-21; First posted 2022-06-24 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: HIV
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Engagement in biosensor wearing (Experimental): A subset of the participants will receive the same interventions, namely the reciprocity messages, personalized feedback, or no prompt (as control condition), using micro-randomization procedure that randomly assign one of the condition in the morning and one of the condition in the evening.
  Interventions: Behavioral: eWrapper-Engagement strategies to facilitate alcohol biosensor wearing

INTERVENTIONS:
Behavioral: eWrapper-Engagement strategies to facilitate alcohol biosensor wearing — We will conduct a 30-day micro-randomized trial (MRT)--a clinical trial design for developing and optimizing mHealth interventions to test which engagement strategy works better, for who, and under what condition. A subset of the participants will be micro-randomized in the morning and in the evening, to either a prompt delivering non-contingent small reward (reciprocity); or a prompt containing feedback on self-monitoring progress based on dynamic self-regulation theories (personalized feedback); or no prompt.

SUMMARY:
In this study, participants will be asked to wear a wrist alcohol biosensor for 30 days and report alcohol use using a ecological momentary assessment (EMA) app. A subset of the sample will be micro-randomized to test two engagement strategies--reciprocity and personalized feedback via the eWrapper app to promote their engagement with the biosensor.

DETAILED DESCRIPTION:
YPLWH (N = 160, 136 after 15% attrition, 18-29 years of age, estimated to include 73% male, 26% female, 1% transgender, 70% racial and ethnic minorities) will be asked to wear a wrist alcohol biosensor (BACtrack Skyn) for 30 days and report their alcohol use using daily ecological momentary assessment (EMA). A subset of the sample will also be micro-randomized twice daily to test two empirically-based engagement strategies - reciprocity and personalized feedback. Data from the 30-day MRT will be used to (a) develop and validate the algorithm for alcohol detection based on Skyn data; and (b) address scientific questions concerning which engagement strategy works best, for whom and under what conditions in terms of facilitating proximal engagement in biosensor wearing. We will also collect alcohol biomarker (i.e., PEth) at 1-month follow up.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and 0 months to 29 years and 11 months
* Currently reside in Florida
* Report having had at least 1 alcoholic drink in the last 30 days
* Able to read and understand English
* Have internet access via smartphone, tablet or computer
* Be diagnosed as HIV positive and;
* Willing to provide informed consent.

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults
* Individuals who are not diagnosed as HIV+
* Prisoners
* Pregnant women

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
Engagement in biosensor wearing | Within 12 hours after prompted engagement strategy
  For the whole sample, it is an observational study, so the outcome is just percentage of biosensor wearing during the 30 day period.
  For the subset who also go through MRT for engagement strategies, we will test the effect of each strategy using % time wearing the sensor in the next 12 hours as the proximal outcome. We hypothesize that the engagement strategies will be better than no prompt and that reciprocity will have an advantage over personalized feedback as it requires less cognitive processing.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - The University of Florida, Gainesville, Florida
  - Florida State University, Tallahassee, Florida
  - The University of Michigan, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Carpenter SM, Case S, Lustria MLA, Marks LR, Yu Q, MacDonell K, Naar S, Wang Y. Feasibility of mHealth Strategies to Promote Use of Wrist-Worn Alcohol Biosensors Among Young Adults With HIV: Protocol for the Engage Microrandomized Trial. JMIR Res Protoc. 2025 Nov 12;14:e69966. doi: 10.2196/69966. PMID 41223419

DOCUMENTS (1):
  • Informed Consent Form (2024-09-04): https://cdn.clinicaltrials.gov/large-docs/55/NCT05431855/ICF_000.pdf